CLINICAL TRIAL: NCT02426918
Title: A Phase 2, Randomized, Double-Blind, Multicenter Study of Safety, Tolerability, and Efficacy of Debio 1450 vs Vancomycin (IV)/Linezolid (Oral) in the Treatment of Acute Bacterial Skin and Skin Structure Infections (ABSSSI) Due to Staphylococcus Sensitive or Resistant to Methicillin
Brief Title: Study of Debio 1450 for Bacterial Skin Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Debio 1450-ABSSSI-201; 218187 (Other: CRO)
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — afabicin; Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Debio 1450 320/480 mg (Experimental): After 2 doses of Debio 1450 IV (intravenous) therapy, the Debio 1450 320/480 mg daily dose group receives 240 mg Debio 1450 Oral + Linezolid Placebo twice daily (BID).
  Interventions: Drug: Debio 1450 IV; Drug: Debio 1450 Oral; Drug: Linezolid Placebo
- Debio 1450 160/240 mg (Experimental): After 2 doses of Debio 1450 IV therapy, the Debio 1450 160/240 mg daily dose group receives 120 mg Debio 1450 Oral + Debio 1450 Oral Placebo + Linezolid Placebo BID.
  Interventions: Drug: Debio 1450 IV; Drug: Debio 1450 Oral; Drug: Debio 1450 Oral Placebo; Drug: Linezolid Placebo
- Placebo (Placebo Comparator): After 2 doses of Vancomycin IV, the Placebo comparator group receives Debio 1450 Oral Placebo + Linezolid 600 mg BID.
  Interventions: Drug: Linezolid; Drug: Debio 1450 Oral Placebo; Drug: Vancomycin IV

INTERVENTIONS:
Drug: Debio 1450 IV — Intravenous (IV) form of Debio 1450 will be supplied in vials containing 50 mg of active pharmaceutical ingredient (API). Intravenous infusions of Debio 1450 (160 mg and 80 mg) will be administered over a 2-hour period BID every 12 hours within a 2-hour window (12 ± 2 hours).
  Arms: Debio 1450 160/240 mg; Debio 1450 320/480 mg
Drug: Debio 1450 Oral — Oral forms of Debio 1450 will be provided as white, opaque, hard gelatin capsules containing 50 mg drug substance (equivalent to 40 mg of Debio 1450).
  Arms: Debio 1450 160/240 mg; Debio 1450 320/480 mg
Drug: Linezolid — Linezolid for oral administration will be provided as 600-mg film-coated compressed tablets.
  Arms: Placebo
Drug: Debio 1450 Oral Placebo — Debio 1450 placebo will be supplied as white, opaque, hard gelatin capsules.
  Arms: Debio 1450 160/240 mg; Placebo
Drug: Linezolid Placebo — Linezolid placebo will be supplied as film-coated compressed tablets.
  Arms: Debio 1450 160/240 mg; Debio 1450 320/480 mg
Drug: Vancomycin IV — Vancomycin will be administered BID every 12 ± 2 hours at doses of 1 g or 15 mg/kg as specified in local protocols, with the infusion rate adjusted to 2 hours.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 2 different doses of intravenous and oral Debio 1450 compared with intravenous vancomycin and oral linezolid in the treatment of patients with staphylococcal ABSSSI.

ELIGIBILITY:
Inclusion Criteria:

* Has clinically documented infection of the skin or skin structure suspected or documented to be caused by a staphylococcal pathogen
* Meets other protocol-specified criteria for qualification and contraception
* Is willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related to food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding);
  3. the analysis of results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Dream Team Clinical Research, LLC, Anaheim, California
  - Physician Alliance Research Center, Anaheim, California
  - Southbay Pharma Research, Buena Park, California
  - eStudySite - Chula Vista, Chula Vista, California
  - eStudySite - La Mesa, La Mesa, California
  - Long Beach Clinical Trials LLC, Long Beach, California
  - Alliance Research, Long Beach, California
  - Central Valley Research, LLC, Modesto, California
  - eStudySite - Oceanside, Oceanside, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Shands Burn Center at the University of Florida, Gainesville, Florida
  - Central Florida Internists, Orlando, Florida
  - Triple O Research Institute, West Palm Beach, Florida
  - Columbus Regional Research, Columbus, Georgia
  - Beaumont Infectious Disease Services, Royal Oak, Michigan
  - Mercury Street Medical Group PLLC, Butte, Montana
  - eStudySite - Las Vegas, Las Vegas, Nevada
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - ID Clinical Research, Ltd., Toledo, Ohio
  - East Montgomery County Clinic, Houston, Texas
  - Tidwell Medical Center, Splendora, Texas

REFERENCES:
- [Derived] Wittke F, Vincent C, Chen J, Heller B, Kabler H, Overcash JS, Leylavergne F, Dieppois G. Afabicin, a First-in-Class Antistaphylococcal Antibiotic, in the Treatment of Acute Bacterial Skin and Skin Structure Infections: Clinical Noninferiority to Vancomycin/Linezolid. Antimicrob Agents Chemother. 2020 Sep 21;64(10):e00250-20. doi: 10.1128/AAC.00250-20. Print 2020 Sep 21. PMID 32747361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study in the United States, from 14 May 2015 to 12 September 2016. Of the 505 participants screened, 175 discontinued from the study prior to randomization and 330 were randomized.
Pre-assignment Details: Participants with acute bacterial skin and skin structure infections (ABSSSI) due to Staphylococcus sensitive or resistant to Methicillin were randomized to one of the three treatment arms in a 1:1:1 ratio.
Groups:
- Debio 1450 80 mg (Milligrams)/120 mg BID: Debio 1450 80 mg was administered intravenously twice daily (BID). After 2 doses of Debio 1450 intravenous (IV) therapy, Debio 1450 80 mg/120 mg daily dose group received 120 mg Debio 1450 Oral + 3 dose of Debio 1450 Placebo + Linezolid matching-Placebo BID.
- Debio 1450 160 mg/240 mg BID: Debio 1450 160 mg was administered intravenously BID. After 2 doses of Debio 1450 IV therapy, Debio 1450 160/240 mg daily dose group received 240 mg Debio 1450 Oral + Linezolid matching-Placebo BID.
- Vancomycin/Linezolid BID: Vancomycin was administered intravenously BID at doses of 1 gram (g) or 15 milligrams per kilogram (mg/kg). After 2 doses of Vancomycin IV, Placebo comparator group received Debio 1450 matching oral placebo + Linezolid 600 mg BID.
Period: Overall Study
Arm/Group | Debio 1450 80 mg (Milligrams)/120 mg BID | Debio 1450 160 mg/240 mg BID | Vancomycin/Linezolid BID
Started | 110 | 109 | 111
Safety Population | 110 | 107 | 107
Completed | 93 | 90 | 97
Not Completed | 17 | 19 | 14
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 5 | 4
Not completed — Other | 9 | 11 | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population (ITT) population included all randomized participants.
Groups:
- Debio 1450 80 mg/120 mg BID: Debio 1450 80 mg was administered intravenously BID. After 2 doses of Debio 1450 IV therapy, the Debio 1450 80 mg/120 mg daily dose group received 120 mg Debio 1450 Oral + 3 dose of Debio 1450 Placebo + Linezolid matching-Placebo BID.
- Debio 1450 160 mg/240 mg BID: Debio 1450 160 mg was administered intravenously BID. After 2 doses of Debio 1450 IV therapy, the Debio 1450 160/240 mg daily dose group received 240 mg Debio 1450 Oral + Linezolid matching-Placebo BID.
- Vancomycin/Linezolid BID: Vancomycin was administered intravenously BID at doses of 1 g or 15 mg/kg. After 2 doses of Vancomycin IV, the Placebo comparator group received Debio 1450 matching oral placebo + Linezolid 600 mg BID.
- Total: Total of all reporting groups
Arm/Group | Debio 1450 80 mg/120 mg BID | Debio 1450 160 mg/240 mg BID | Vancomycin/Linezolid BID | Total
Number analyzed (Participants) | 110 | 109 | 111 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (11.71) | 42.8 (11.72) | 44.8 (10.57) | 43.8 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 32 | 103
  Male | 74 | 74 | 79 | 227

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response Rate (ECRR): Percentage of Responders to Treatment at 48 to 72 Hours From Randomization as Assessed by the Investigator
Description: ECRR was defined as the percentage of responders to treatment at 48 to 72 hours from randomization. Responders were the participants who showed greater than or equal to (≥) 20% reduction in area of the primary lesion involving erythema, edema, or induration of the primary ABSSSI lesion (as assessed by the ruler method) at 48 to 72 hours compared to baseline.
Time Frame: At 48 to 72 hours from randomization (Day 4)
Population: Microbiological Intent-to-Treat (mITT) population included all randomized participants who were culture positive for any staphylococcal species considered pathogenic and received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Debio 1450 80 mg/120 mg BID | Debio 1450 160 mg/240 mg BID | Vancomycin/Linezolid BID
Number analyzed (Participants) | 92 | 91 | 101
percentage of participants | 94.6 | 90.1 | 91.1
Statistical Analysis 1: Comparison: Debio 1450 80 mg/120 mg BID vs Vancomycin/Linezolid BID; Treatment difference estimates and 95% CIs are calculated accounting for the randomization strata infection type [cellulitis, noncellulitis] according to a Mantel-Haenszel type risk difference estimator; Test type: Non-Inferiority — Non-inferiority for the low dose was confirmed if the upper bound of the CI was < 15% and if non-inferiority was confirmed for the high dose; Risk Difference (RD) = -4.2, 95% CI 2-sided [-11.42 to 3.00]
Statistical Analysis 2: Comparison: Debio 1450 160 mg/240 mg BID vs Vancomycin/Linezolid BID; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Non-inferiority for the high dose was confirmed if the upper bound of the CI was < 15%; Risk Difference (RD) = 0.0, 95% CI 2-sided [-8.32 to 8.38]

2. Secondary Outcome: Clinical Success Rate: Percentage of Participants Assessed by the Investigator as Responders at 48 to 72 Hours From Randomization, at End of Treatment (EOT) and Short-term Follow-up (STFU)
Description: The Investigator Assessment of Clinical Outcome (IACO) of treatment was assessed for each participant as success or failure at 48 to 72 hours after randomization at EOT and STFU visits. Clinical success was resolution or near resolution of most disease-specific signs and symptoms and no new signs, symptoms, or complications attributable to ABSSSI such that no further antibiotic therapy is required for treatment of original site of infection. Clinical failure was requirement for additional antibiotic therapy for treatment of the original site of infection or incision and drainage of ABSSSI site that was not both anticipated and completed within a 48- to 72-hour window following randomization, or unplanned major surgical intervention required due to failure of study medication or development of osteomyelitis after baseline. Participants who met both success criteria and none of failure criteria were considered as a clinical success for IACO.
Time Frame: 48 to 72 hours after randomization (Day 4), EOT (Day 12) and STFU (Day 19)
Population: mITT population included all randomized participants who were culture positive for any staphylococcal species considered pathogenic and received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Debio 1450 80 mg/120 mg BID | Debio 1450 160 mg/240 mg BID | Vancomycin/Linezolid BID
Number analyzed (Participants) | 92 | 91 | 101
percentage of participants
  48 to 72 hours after randomization | 83.7 | 81.3 | 86.1
  EOT | 92.4 | 87.9 | 92.1
  STFU | 84.8 | 83.5 | 92.1

3. Secondary Outcome: Clinical Success Rate: Percentage of Participants Assessed by the Sponsor as Responders After 7 to 10 Days of Treatment at EOT and STFU
Description: The Sponsor's Assessment of Clinical Outcome was obtained at EOT and STFU visits based on IACO and additional criteria. Sponsor assessed participants as clinical failure if they required non-study or rescue antibiotics due to lack of efficacy after at least 48 hours from randomization or experienced drug-related serious adverse events (SAEs) or discontinuation of study medication for drug-related AEs or required antibiotic therapy for longer than 10 days or had the need for unplanned surgical intervention >48 hours after randomization. As per IACO, clinical success was resolution or near resolution of most disease-specific signs and symptoms and no new signs, symptoms or complications. Clinical failure was requirement for additional antibiotic therapy or incision and drainage of ABSSSI site or unplanned major surgical intervention or development of osteomyelitis.
Time Frame: EOT (Day 12) and STFU (Day 19)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Debio 1450 80 mg/120 mg BID | Debio 1450 160 mg/240 mg BID | Vancomycin/Linezolid BID
Number analyzed (Participants) | 92 | 91 | 101
percentage of participants
  EOT | 89.1 | 86.8 | 90.1
  STFU | 81.5 | 81.3 | 90.1

4. Secondary Outcome: Percentage of Participants With a Composite Assessment of Clinical Outcome (CACO) of Success
Description: CACO of treatment was determined as a combined outcome of early response to treatment (at 48 to 72 hours from randomization) and IACO at the STFU visit. Participants had a CACO of success if they met both of the following criteria: An early response to treatment (at 48 to 72 hours from randomization) (ECR = responder) and a clinical outcome of success at the STFU visit (7 to 14 days after EOT) based on IACO (IACO = success).
Time Frame: 48 to 72 hours after randomization (Day 4) and STFU (Day 19)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Debio 1450 80 mg/120 mg BID | Debio 1450 160 mg/240 mg BID | Vancomycin/Linezolid BID
Number analyzed (Participants) | 92 | 91 | 101
percentage of participants | 83.7 | 81.3 | 88.1

5. Secondary Outcome: Percentage of Participants Who Showed Microbiological Evidence of Cure 48 to 72 Hours From Randomization, EOT, and STFU
Description: The microbiological outcome was assessed by the sponsor at 48 to 72 hours from randomization, EOT and STFU. It was based on blood and skin lesion identification results from baseline samples and skin lesion identification results from baseline samples and skin lesion identification results from follow-up samples as well as on, molecular typing results, and the IACO. Microbiological eradication rate was defined as proportion of participants with 'Documented Eradication' (absence of baseline pathogen(s) in follow-up cultures of the original site of infection.) or 'Presumed Eradication' (no material available for culture and an IACO of 'Success') in relation to the total number of participants in the respective treatment group.
Time Frame: 48 to 72 hours after randomization (Day 4), EOT (Day 12) and STFU (Day 19)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Debio 1450 80 mg/120 mg BID | Debio 1450 160 mg/240 mg BID | Vancomycin/Linezolid BID
Number analyzed (Participants) | 92 | 91 | 101
percentage of participants
  48 to 72 hours after randomization | 72.8 | 69.2 | 75.2
  EOT | 92.4 | 86.8 | 91.1
  STFU | 84.8 | 83.5 | 91.1

ADVERSE EVENTS:
Time Frame: 21 days after EOT (Day 33)
Description: Safety population included all participants who received at least one dose of study medication.
Arm/Group | Debio 1450 80 mg/120 mg BID | Debio 1450 160 mg/240 mg BID | Vancomycin/Linezolid BID
Serious Adverse Events (participants affected / at risk) | 2/110 | 1/107 | 1/107
Other Adverse Events (participants affected / at risk) | 18/110 | 29/107 | 20/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Debio 1450 80 mg/120 mg BID (N=110) | Debio 1450 160 mg/240 mg BID (N=107) | Vancomycin/Linezolid BID (N=107)
Cellulitis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 2 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Debio 1450 80 mg/120 mg BID (N=110) | Debio 1450 160 mg/240 mg BID (N=107) | Vancomycin/Linezolid BID (N=107)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 6
Nausea (Gastrointestinal disorders) | 7 | 9 | 7
Vomiting (Gastrointestinal disorders) | 1 | 6 | 2
Abscess (Infections and infestations) | 3 | 6 | 0
Headache (Nervous system disorders) | 10 | 18 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or scientific communication related to this study can only take place once the agreement between the Sponsor and the Investigator has been reached.